CLINICAL TRIAL: NCT06039891
Title: A Single-arm, Single-center, Prospective, Phase II Study of Nimotuzumab, Tislelizumab Plus Radiotherapy for Recurrent and Metastatic Cervical Cancer
Brief Title: Nimotuzumab Plus Tislelizumab for Recurrent and Metastatic Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lei Li, chief physician, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K4391
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab; tislelizumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab, Tislelizumab group (Experimental): Subjects will receive Nimotuzumab 400 mg/time, intravenous injection, qw; Tislelizumab 200 mg/time, q3w until disease progression, intolerable toxicity, or 24 months of medication
  Interventions: Drug: Nimotuzumab、Tislelizumab

INTERVENTIONS:
Drug: Nimotuzumab、Tislelizumab — Subjects will receive Nimotuzumab 400 mg/time, intravenous injection, qw; Tislelizumab 200 mg/time, q3w until disease progression, intolerable toxicity, or 24 months of medication
  Other Names: Nimotuzumab, Tislelizumab plus radiotherapy

SUMMARY:
Patients with recurrent or metastatic cervical cancer have very poor prognosis. For eligible patients, radiotherapy remains the choice, which has the most effective impact on the survival periods. Epidermal growth factor receptor (EGFR) is overexpressed in cervical cancer cells, anti-EGFR therapy maybe an ideal target for the treatment of cervical cancer. This study aims to discover the progression-free survival of combination therapy with nimotuzumab (an anti-epidermal growth factor receptor [EGFR] IgG1 humanized monoclonal antibody) 、Tislelizumab and radiotherapy in recurrent or metastatic uterine cervical squamous carcinoma in a single-arm, open, phase 2 clinical trial.

DETAILED DESCRIPTION:
Nimotuzumab, is a humanized antibody recognizing with high affinity the epidermal growthfactor (EGF-R)，has shown promising efficacy and tolerable toxicity in the cervical cancer. In this study, patients with recurrent or metastatic cervical cancer, will be included in this study according to the prescribed criteria in the protocal. Nimotuzumab 400 mg/time, intravenous injection, qw; Tislelizumab 200 mg/time, q3w until disease progression, intolerable toxicity, or 24 months of medication. Assess objective response rate; progression-free survival; median overall survival and safety ( adverse event).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18；
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2；
3. Have recurrent, or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix；
4. Oligometastases and Oligo-recurrence( number of metastatic organs ≤3, and the total number of metastases ≤5), with indications for radiotherapy, and which has not been treated with systemic chemotherapy；
5. At least one measurable lesion defined by Response Evaluation Criteria in Solid Tumors (RECIST) guideline 1.1；
6. Anticipative survival period of 3 months or more；
7. Have adequate organ function as indicated by the following laboratory values： (1) Hematological：Absolute neutrophil count (ANC)≥1.5×109/L；Platelets(PLT)≥90×109/L；Hemoglobin(Hb)≥90 g/L； (2) Hepatic：Serum total bilirubin (TBIL)≤2.5×ULN；ALT 和 AST≤2×ULN； (3) Renal:BUN 和 Cr ≤ 1.5×ULN；
8. Cardiac ultrasound：LVEF≥50%；
9. A WOCBP who has a positive blood pregnancy test within 72 hours prior to randomization（Postmenopausal women who have had amenorrhea for at least 12 months are considered infertile, and women who are known to have received Tubal ligation do not require a pregnancy test）；
10. For subjects who were not menopausal or had not undergone surgical sterilization, consent to abstinence or use of an effective contraceptive method was given during treatment and at least 5 months after the last administration of the drug during study treatment;
11. Volunteer to join the study, sign informed consent, have good compliance and willing to cooperate with the follow-up.

Exclusion Criteria:

1. Patients who have received prior therapy with an anti-EGFR an anti-PD-1, anti-PD-L1 agent; Has a contraindication or hypersensitivity to Macromolecular protein preparationsany and component of Nimotuzumab and Tislelizumab
2. Other malignancies diagnosed within 5 years before the first dose, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin and papillary thyroid carcinoma;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy， prior therapy with other targeted therapy and any anti-vascular endothelial growth factor (VEGF) drug. Other anti-tumor treatments not included in this trial protocol；
4. Patients who are pregnant or nursing. Patients of childbearing potential must agree to use contraceptive measures during study therapy and for at least five months after completion of this study.
5. Patients with recto-vaginal fistula,vesicovaginal fistula, uncontrolled vaginal bleeding and no underlying process leading to fistula；
6. Major surgical procedure unrelated to cervical cancer,and has not recovered adequately from toxicity and/or complications from surgery within 4 weeks before enrollment；
7. Has a known history of human immunodeficiency virus (HIV) infection,or has other acquired, congenital immunodeficiency disease, or has a history of organ transplantation；
8. Uncontrolled hypertension , cardiac arrhythmia and pulmonary disease.Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg]reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
9. Has known active Central Nervous System (CNS)metastases and/or carcinomatous meningitis. Participants with known brain metastases may participate provided that the brain metastases have been previously treated (except with chemotherapy) and are radiographically stable more than 2 weeks. Known brain metastases are considered active, if any of the following criteria are: There were measurable lesions outside the central nervous system, no metastases to meninges, midbrain, pons, cerebellum, medulla oblongata or spinal cord, no previous history of intracranial hemorrhage, and steroid therapy was discontinued 14 days before the first dose of study drug.
10. Patients with clinical signs or fluids of pleural effusion, ascites, or pericardial effusion requiring drainage (required or not significantly increased within 3 days of discontinuation of drainage) may be eligible;
11. Any previous arterial thrombosis, thrombosis, or ischaemia, such as myocardial infarction, unstable angina, cerebrovascular accident, etc., occurred in the previous 6 months.A history of deep venous thrombosis or any other serious thromboembolism (implanted venous port or catheter-derived thrombosis, superficial venous thrombosis, or thromboembolic stability after conventional therapy were not considered as serious" thromboembolism" during the first 3 months of enrollment";
12. Cancer thrombus in the portal vein involves both the main and right branches of the portal vein, or both the main and the superior mesenteric and inferior vena cava thrombus; the superior vena cava thrombus and the superior vena cava syndrome;
13. Tumour involvement of vital peripheral organs or vessels (such as the great vessels of the mediastinum, superior vena cava, inferior vena cava, abdominal aorta, iliac vessels, trachea, esophagus, etc.) or risk of esophageal-tracheal or esophageal pleural fistula;
14. History of interstitial pneumonia, pharmacologic pneumonia, radiation pneumonia, idiopathic pneumonia, or active pneumonia;
15. Severe infection in active state or under clinical control.Severe infections occurred within 4 weeks before the first dose, including but not limited to hospitalization for infection, bacteremia, or complications of severe pneumonia.
16. Inability to perform internal exposure therapy by the Investigator's assessment；
17. Patients who do not understand the requirements of the trial or may not comply with them.
18. Participants were identified as having any medical, psychiatric, or other condition or condition that may adversely affect their safety or the reliability of study data.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | one year
  Progression-free survival is defined as the time from the start of treatment with caldonirimab and nimotuzumab until the first documentation of disease progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Objective response rate (ORR) | one year
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1
Median Overall survival（mOS） | three years
  Overall survival from the start of study to the disease progression
Adverse events (AEs) | three years
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment